CLINICAL TRIAL: NCT07131995
Title: Formative Usability Testing Study of a Novel Medical Device for Peritoneal Dialysis (WEAKID)
Acronym: WEAKID
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Hospital Universitario La Paz (Other); Azienda Unita' Sanitaria Locale Di Modena (Other)
Responsible Party: Principal Investigator, Karin G.F. Gerritsen, Principal Investigator, UMC Utrecht
Other Study IDs: 21/616
Record Dates: First submitted 2025-07-15; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses: Nurses, aged 18 years or older, and having >1 years of professional experience with PD.
- Patients: Patients, aged 18 years or older, having a clinical diagnosis of ESRD and any treatment experience with PD, either current or in the past.

SUMMARY:
This study aimed to formatively test the usability of the WEarable Artificial KIDney (WEAKID) for peritoneal dialysis (PD) in the device's intended user populations (i.e., nurses and patients).

DETAILED DESCRIPTION:
End stage renal disease is a growing health problem worldwide, with a growing number of patients requiring a kidney transplantation. Recent years have seen the development of multiple novel devices for both hemodialysis and peritoneal dialysis (PD), one of these devices being the WEarable Artificial KIDney (WEAKID) for PD. WEAKID uses both sorbent technology and continuous flow PD to improve dialysis efficacy. Here, we present the results of a formative usability testing study of WEAKID among nurses and patients. We included 14 participants (n=6 nurses, n=8 patients) in three participating centres (Modena University Hospital, Italy; La Paz University Hospital Madrid, Spain; University Medical Center Utrecht, the Netherlands). Participants were asked to perform basic operational procedures with the device according to a usability task list. Their performance was observed and use errors were noted. Furthermore, participants were asked for feedback, both verbally and by means of completing the system usability scale (SUS), reflecting perceived usability on a scale from 0 (worst) to 100 (best). In total, 22 use errors occurred, 10 in nurses and 12 in patients. The mean SUS score was 70 (range 57.5 - 85) for nurses, and 71.9 (range 55 - 87.5) for patients. Despite the slightly above-average perceived usability of the device's current design stage, participants made a lot of suggestions for improvements, and indeed, usability must be improved to make the device ready for market introduction.

ELIGIBILITY:
Inclusion Criteria:

* Nurses: aged 18 years or older, >1 years of professional experience with PD.
* Patients: aged 18 years or older, clinical diagnosis of ESRD, any treatment experience with PD, either current or in the past.

Exclusion Criteria:

* Nurses: none.
* Patients: severe physical and/or cognitive impairment, as judged by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants represented two populations of intended users of the device, namely nurses and patients. The sample sizes were set at 6 (nurses) and 8 (patients). Prior work on the sample sizes of formative usability testing has shown that these sample sizes suffice to identify the most important design issues.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Use errors | During the procedure (usability test)
  The number and percentages of incorrect actions during task performance. Reported per participant and for the total group.

SECONDARY OUTCOMES:
Completion rate | During the procedure (usability test)
  The number and percentages of tasks successfully completed during task performance. Reported per participant and for the total group.
Perceived usability | Immediately after the procedure (usability test)
  Participants' perceived usability of the device using the 10-item System Usability Scale (0-100 scale). Scores were reported per participant and for the total group.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No
Privacy-sensitive information